CLINICAL TRIAL: NCT01616693
Title: Supplementation With Zinc and/or Probiotics to Enhance the Immune Response of Oral Rotavirus and Polio Vaccines in Indian Infants
Brief Title: Zinc and/or Probiotic Supplementation of Rotavirus and Oral Polio Virus Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Christian Medical College, Vellore, India (Other); Ministry of Science and Technology, India (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CMC ZP 2012; PATH HS-658
Record Dates: First submitted 2012-06-06; First posted 2012-06-12 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Immunity to Oral Rotavirus Vaccine; Immunity to Oral Polio Vaccine; Shedding of Oral Rotavirus Vaccine
Keywords: rotavirus; polio; zinc supplement; probiotic supplement; rotavirus vaccine shedding
MeSH Terms: conditions — Poliomyelitis | interventions — Probiotics; Zinc; Rotavirus Vaccines; RIX4414 vaccine; Poliovirus Vaccine, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Zinc and probiotic (Experimental): Received daily zinc and probiotic supplements, in addition to rotavirus vaccine and trivalent oral polio vaccines.
  Interventions: Dietary Supplement: Probiotic; Dietary Supplement: Zinc; Biological: Rotavirus vaccine; Biological: Oral polio vaccine
- Zinc alone (Active Comparator): Received daily zinc and probiotic placebo supplement, in addition to rotavirus vaccine and trivalent oral polio vaccine.
  Interventions: Dietary Supplement: Zinc; Dietary Supplement: Probiotic placebo; Biological: Rotavirus vaccine; Biological: Oral polio vaccine
- Probiotic alone (Active Comparator): Received daily zinc placebo and probiotic supplement, in addition to rotavirus vaccine and trivalent oral polio vaccine.
  Interventions: Dietary Supplement: Probiotic; Dietary Supplement: Zinc placebo; Biological: Rotavirus vaccine; Biological: Oral polio vaccine
- Placebo (Placebo Comparator): Received daily zinc placebo and probiotic placebo, in addition to rotavirus vaccine and trivalent oral polio vaccine.
  Interventions: Dietary Supplement: Probiotic placebo; Dietary Supplement: Zinc placebo; Biological: Rotavirus vaccine; Biological: Oral polio vaccine

INTERVENTIONS:
Dietary Supplement: Probiotic — A capsule that contains at least 1 x 10^9 Lactobacillus rhamnosus GG organisms per capsule. The contents of this capsule were given once daily orally.
  Other Names: Culturelle
  Arms: Probiotic alone; Zinc and probiotic
Dietary Supplement: Zinc — Zinc sulphate syrup is zinc sulphate heptahydrate (concentration 1mg/ml). 5 ml of this suspension was given once daily orally.
  Arms: Zinc alone; Zinc and probiotic
Dietary Supplement: Probiotic placebo — The probiotic placebo was manufactured by the same company that manufactured the probiotic and contained inulin powder but no Lactobacillus rhamnosus GG. The contents of the capsule were given once daily orally.
  Arms: Placebo; Zinc alone
Dietary Supplement: Zinc placebo — The zinc placebo excluded the zinc sulphate but contained lactose and was diluted to match the taste. 5 ml of this suspension was given orally once daily.
  Arms: Placebo; Probiotic alone
Biological: Rotavirus vaccine — 1 ml Rotarix®, a lyophilized human rotavirus vaccine reconstituted with calcium carbonate buffer provided orally at 6 and 10 weeks.
  Other Names: Rotarix®
Biological: Oral polio vaccine — A liquid trivalent polio vaccine provided orally at 6 and 10 weeks.
  Other Names: Biopolio®

SUMMARY:
Background: Strategies are needed to improve oral rotavirus vaccine (RV), which provides suboptimal protection in developing countries. Probiotics and zinc supplementation could improve RV immunogenicity by altering the intestinal microbiota and immune function.

This study enrolled infants 5 weeks old living in urban Vellore, India to assess the effects of daily zinc (5 mg), probiotic (1010 Lactobacillus rhamnosus GG) or placebo on the immunogenicity of two doses of RV (Rotarix,GlaxoSmithKline Biologicals) given at 6 and 10 weeks of age. Probiotics and zinc (or placebo) were provided for six weeks. A single dose of test product was administered daily one week prior to first study dose of rotavirus and polio vaccines through 1 week following second study dose of rotavirus and polio vaccines.

DETAILED DESCRIPTION:
Co- Primary objectives:

1. To evaluate the serologic immune response to rotavirus vaccine (sero-conversion or four-fold rise in rotavirus immunoglobulin A (IgA) antibodies) among Indian infants receiving zinc supplementation given daily for a week prior to the administration of the first dose through a week following the second dose of oral rotavirus vaccine compared to those receiving a zinc placebo.
2. To evaluate the serologic immune response to rotavirus vaccine (sero-conversion or four-fold rise in rotavirus IgA antibodies) among Indian infants receiving probiotic supplementation given daily for a week prior to the administration of the first dose through a week following the second dose of oral rotavirus vaccine compared to those receiving a probiotic placebo.

ELIGIBILITY:
Inclusion Criteria:

* Infants 35-41 days old
* Live in area under surveillance
* Current weight ≥3.2 kg
* No syndromic evidence of immunocompromise as determined by medical doctor
* No prior illness requiring hospitalization
* No current medical condition as determined by medical doctor which precludes study involvement
* Available for follow up for duration of study (through approximately 14 weeks of age)
* Parents/guardians of infant are able to understand and follow study procedures and agree to participate in the study by providing signed informed consent

Exclusion Criteria:

* Child has history of atopic symptoms
* Child has a known digestive system defect
* Child has history of chronic diarrhea
* Child has major congenital anomalies
* Child has received a prior dose of rotavirus vaccine
* Child has received a prior dose of polio vaccine (beyond the birth dose)

Ages: 5 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 620 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gagandeep Kang, MD, PhD, Principal Investigator — Christian Medical Center, Vellore, India
Locations (1):
- Christian Medical Center, Vellore, Vellore, Tamil Nadu, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants for this study lived in the area surrounding the Christian Medical College (CMC) in the town of Vellore, Tamil Nadu, India. Parents were contacted through the existing Demographic Surveillance System shortly after the child's birth. Procedures were conducted in the Chinallapuram Field Clinic.
Groups:
- Zinc Alone: Received daily zinc and probiotic placebo supplement, in addition to rotavirus vaccine and trivalent oral polio vaccine.
  Zinc: Zinc sulphate syrup is zinc sulphate heptahydrate (concentration 1mg/ml). 5 ml of this suspension was given once daily orally.
  Probiotic placebo: The probiotic placebo was manufactured by the same company that manufactured the probiotic and contained inulin powder but no LGG. The contents of the capsule were given once daily orally.
  Rotavirus vaccine: 1 ml Rotarix®, a lyophilized human rotavirus vaccine reconstituted with calcium carbonate buffer provided orally at 6 and 10 weeks.
  Oral polio vaccine: A liquid trivalent polio vaccine provided orally at 6 and 10 weeks.
- Placebo: Received daily zinc placebo and probiotic supplement, in addition to rotavirus vaccine and trivalent oral polio vaccine.
  Probiotic placebo: The probiotic placebo was manufactured by the same company that manufactured the probiotic and contained inulin powder but no LGG. The contents of the capsule were given once daily orally.
  Zinc placebo: The zinc placebo excluded the zinc sulphate but contained lactose and was diluted to match the taste. 5 ml of this suspension was given orally once daily.
  Rotavirus vaccine: 1 ml Rotarix®, a lyophilized human rotavirus vaccine reconstituted with calcium carbonate buffer provided orally at 6 and 10 weeks.
  Oral polio vaccine: A liquid trivalent polio vaccine provided orally at 6 and 10 weeks.
Period: Evaluated for Safety
Arm/Group | Zinc and Probiotic | Zinc Alone | Probiotic Alone | Placebo
Started | 155 | 155 | 155 | 155
Completed | 154 | 155 | 154 | 155
Not Completed | 1 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0
Period: Received Both Vaccines
Arm/Group | Zinc and Probiotic | Zinc Alone | Probiotic Alone | Placebo
Started | 154 | 155 | 154 | 155
Completed | 141 | 145 | 142 | 136
Not Completed | 13 | 10 | 12 | 19
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 7 | 8 | 15
Not completed — Lost to Follow-up | 4 | 3 | 4 | 4
Period: Blood Analyzed for Immunogenicity
Arm/Group | Zinc and Probiotic | Zinc Alone | Probiotic Alone | Placebo
Started | 141 | 145 | 142 | 136
Completed | 137 | 143 | 136 | 135
Not Completed | 4 | 2 | 6 | 1
Not completed — Protocol Violation | 4 | 2 | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zinc and Probiotic | Zinc Alone | Probiotic Alone | Placebo | Total
Number analyzed (Participants) | 155 | 155 | 155 | 155 | 620
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 5.1 (.3) | 5.1 (.3) | 5.1 (.3) | 5.2 (.3) | 5.1 (.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 87 | 80 | 84 | 326
  Male | 80 | 68 | 75 | 71 | 294
Region of Enrollment [Number; unit: participants]
  India | 155 | 155 | 155 | 155 | 620
Religion [Count of Participants; unit: Participants]
  Hindu | 99 | 96 | 116 | 104 | 415
  Christian | 5 | 10 | 5 | 6 | 26
  Muslim | 51 | 49 | 34 | 45 | 179
Type of house [Count of Participants; unit: Participants]
  Permanent (pucca) | 85 | 92 | 93 | 90 | 360
  Mixed | 59 | 47 | 52 | 54 | 212
  Temporary | 11 | 16 | 10 | 11 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number/Percentage of Subjects With Immune Response to Rotavirus Vaccine
Description: Defined as an increase in serum anti-rotavirus (RV) VP6 IgA antibodies consistent with seroconversion (detection of serum anti-RV VP6 immunoglobulin A (IgA) antibodies at a concentration ≥20 U/ml in a previously seronegative individual) or a fourfold rise in anti-RV VP6 IgA antibodies between baseline and 14 weeks of age.
  Pre-vaccination blood samples were taken when the subject received the first dose of rotavirus vaccine (when the subject was 6 weeks of age); post-vaccination blood samples were taken 4 weeks after the second dose of rotavirus vaccine was administered (14 weeks of age).
Time Frame: from first dose of rotavirus vaccine to 4 weeks after last dose of vaccine
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Received daily zinc placebo and probiotic placebo, in addition to rotavirus vaccine and trivalent oral polio vaccine.
  Probiotic placebo: The probiotic placebo was manufactured by the same company that manufactured the probiotic and contained inulin powder but no LGG. The contents of the capsule were given once daily orally.
  Zinc placebo: The zinc placebo excluded the zinc sulphate but contained lactose and was diluted to match the taste. 5 ml of this suspension was given orally once daily.
  Rotavirus vaccine: 1 ml Rotarix®, a lyophilized human rotavirus vaccine reconstituted with calcium carbonate buffer provided orally at 6 and 10 weeks.
  Oral polio vaccine: A liquid trivalent polio vaccine provided orally at 6 and 10 weeks.
- Zinc: All subjects receiving zinc supplementation (zinc and probiotic; zinc and probiotic placebo groups)
- No Zinc: All subjects receiving zinc placebo (group receiving zinc placebo and probiotic, combined with group receiving zinc placebo and probiotic placebo)
- Probiotic: All subjects receiving probiotic supplementation (zinc and probiotic; zinc placebo and probiotic)
- No Probiotic: All subjects receiving probiotic placebo (zinc and probiotic placebo; zinc placebo and probiotic placebo)
Arm/Group | Zinc and Probiotic | Zinc Alone | Probiotic Alone | Placebo | Zinc | No Zinc | Probiotic | No Probiotic
Number analyzed (Participants) | 137 | 143 | 136 | 135 | 280 | 271 | 273 | 278
Participants
  Seroconversion | 54 | 40 | 42 | 37 | 94 | 79 | 96 | 77
  No seroconversion | 83 | 103 | 94 | 98 | 186 | 192 | 177 | 201
Statistical Analysis 1: Comparison: Zinc vs No Zinc; Test type: Superiority; Difference in seroconversion proportion = 4.4, 97.5% CI 2-sided [-4.4 to 13.2]
Statistical Analysis 2: Comparison: Probiotic vs No Probiotic; Test type: Superiority; Difference in seroconversion proportion = 7.5, 95% CI 2-sided [-1.4 to 16.2]
Statistical Analysis 3: Comparison: Zinc and Probiotic vs Placebo; Test type: Superiority; Difference in seroconversion proportion = 12.0, 95% CI 2-sided [.8 to 22.8]

2. Primary Outcome: Geometric Mean Concentration of Rotavirus-specific IgA
Description: Pre-vaccination blood samples were taken when the subject received the first dose of rotavirus vaccine (when the subject was 6 weeks of age); post-vaccination blood samples were taken 4 weeks after the second dose of rotavirus was administered (14 weeks of age).
  Pre-vaccination blood samples were taken when the subject received the first dose of rotavirus vaccine (when the subject was 6 weeks of age); post-vaccination blood samples were taken 4 weeks after the second dose of rotavirus vaccine was administered (14 weeks of age).
Time Frame: from first dose of rotavirus vaccine to 4 weeks after last dose of vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Zinc and Probiotic | Zinc Alone | Probiotic Alone | Placebo | Zinc | No Zinc | Probiotic | No Probiotic
Number analyzed (Participants) | 137 | 143 | 136 | 135 | 280 | 271 | 273 | 278
titer
  Pre-vaccination | 9.3 [7.5 to 11.6] | 10.8 [8.4 to 13.9] | 11.3 [9.0 to 14.2] | 12.2 [9.5 to 15.7] | 10.0 [8.5 to 11.8] | 11.7 [9.9 to 13.9] | 10.2 [8.7 to 12.0] | 11.5 [9.6 to 13.7]
  Post-vaccination | 23.4 [17.5 to 31.3] | 23.9 [17.8 to 32.1] | 25.4 [19.2 to 33.6] | 26.0 [19.3 to 34.9] | 23.7 [19.3 to 29.1] | 25.7 [21.0 to 31.4] | 24.4 [19.9 to 29.8] | 24.9 [20.3 to 30.6]

3. Secondary Outcome: Number/Percentage of Subjects With Immune Response to Trivalent Oral Poliovirus Vaccine (OPV)
Description: A serologic immune response to OPV is defined as a neutralizing antibody titer to polio virus subtype 3 greater than or equal to 1:8 at 14 weeks of age. This antigen will be used as a conservative estimate because it gives the lowest immune response of all three polio antigens.
  Pre-vaccination blood samples were taken when the subject received the first dose of OPV vaccine (when the subject was 6 weeks of age); post-vaccination blood samples were taken 4 weeks after the second dose of OPV was administered (14 weeks of age).
Time Frame: from first dose of OPV to 4 weeks after last dose of OPV
Measure: Count of Participants; unit: Participants
Arm/Group | Zinc and Probiotic | Zinc Alone | Probiotic Alone | Placebo | Zinc | No Zinc | Probiotic | No Probiotic
Number analyzed (Participants) | 137 | 143 | 136 | 135 | 280 | 271 | 273 | 278
Participants
  Seroconversion | 120 | 129 | 117 | 121 | 249 | 238 | 237 | 250
  No seroconversion | 17 | 14 | 19 | 14 | 31 | 33 | 36 | 28
Statistical Analysis 1: Comparison: Zinc vs No Zinc; Test type: Superiority; Mean Difference (Net) = 1.1, 95% CI 2-sided [-4.3 to 6.6]
Statistical Analysis 2: Comparison: Probiotic vs No Probiotic; Test type: Superiority; Mean Difference (Net) = -3.1, 95% CI 2-sided [-8.6 to 2.3]
Statistical Analysis 3: Comparison: Zinc and Probiotic vs Placebo; Test type: Superiority; Mean Difference (Net) = -2.0, 95% CI 2-sided [-9.8 to 5.7]

4. Secondary Outcome: Number/Percentage of Subjects Exhibiting Rotavirus Shedding in Stool After Dose 1
Description: Shedding of rotavirus following vaccination through detection of rotavirus antigen by ELISA and confirmed as vaccine type by Real-time polymerase chain reaction (RT-PCR). Stool samples were collected on Day 0 (i.e., day of vaccination or -1), Day 4 (±1) and Day 7 (-1 to +2) post vaccination.
Time Frame: 0, 4 and/or 7 day post dose 1 of rotavirus vaccine
Population: Subjects who received the vaccination on schedule and had valid stool samples on the days of testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Zinc and Probiotic | Zinc Alone | Probiotic Alone | Placebo | Zinc | No Zinc | Probiotic | No Probiotic
Number analyzed (Participants) | 121 | 119 | 114 | 120 | 240 | 234 | 235 | 239
Participants
  Shedding 4 or 7 days post-vaccination | 1 | 1 | 1 | 2 | 2 | 3 | 2 | 3
  No shedding 4 or 7 days post-vaccination | 120 | 118 | 113 | 118 | 238 | 231 | 233 | 236

5. Secondary Outcome: Number/Percentage of Subjects Exhibiting Rotavirus Shedding in Stool After Dose 2
Description: Shedding of rotavirus following vaccination through detection of rotavirus antigen by ELISA and confirmed as vaccine type by RT-PCR. Stool samples were collected on Day 0 (i.e., day of vaccination or -1), Day 4 (±1) and Day 7 (-1 to +2) post vaccination.
Time Frame: 0, 4 and/or 7 day post dose 2 of rotavirus vaccine
Population: Subjects who received the vaccination on schedule and had valid stool samples on the days of testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Zinc and Probiotic | Zinc Alone | Probiotic Alone | Placebo | Zinc | No Zinc | Probiotic | No Probiotic
Number analyzed (Participants) | 118 | 118 | 114 | 118 | 136 | 132 | 132 | 136
Participants
  Shedding 4 or 7 days post-vaccination | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  No shedding 4 or 7 days post-vaccination | 118 | 118 | 114 | 118 | 136 | 132 | 132 | 136

6. Secondary Outcome: Serious Adverse Events (SAEs)
Description: Field workers documented information on SAEs through the duration of the study during home visits (twice weekly between study clinic visits) or SAEs were documented by study clinicians at the study clinic or hospital. All SAEs occurring at any time during the study were recorded on a SAE Form and were reviewed and evaluated by a study clinician and the local IRB. The relationship of the SAE to study vaccine was evaluated and recorded and reported to the local institutional review board (IRB). All SAEs were followed until satisfactory resolution.
Time Frame: from first day of study to 4 weeks after last dose
Measure: Count of Participants; unit: Participants
Arm/Group | Zinc and Probiotic | Zinc Alone | Probiotic Alone | Placebo
Number analyzed (Participants) | 154 | 155 | 154 | 155
Participants
  Unrelated SAEs | 5 | 3 | 2 | 4
  Related SAEs | 0 | 0 | 0 | 0
  No SAEs | 149 | 152 | 152 | 151

ADVERSE EVENTS:
Time Frame: from first day of study to 4 weeks after last dose (11 weeks)
Description: Field workers documented information on severe adverse events (SAEs) through the duration of the study during home visits (twice weekly between study clinic visits) or SAEs were documented by study clinicians at the study clinic or hospital.
  Adverse events solicited included: diarrhea, vomiting, reported fever, cough, and cold/runny nose. Any other adverse event that was not considered an SAE was documented as "any other illness".
Arm/Group | Zinc and Probiotic | Zinc Alone | Probiotic Alone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/155 | 0/154 | 0/155
Serious Adverse Events (participants affected / at risk) | 5/154 | 3/155 | 2/154 | 4/155
Other Adverse Events (participants affected / at risk) | 149/154 | 152/155 | 148/154 | 146/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zinc and Probiotic (N=154) | Zinc Alone (N=155) | Probiotic Alone (N=154) | Placebo (N=155)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 3
Meningitis (Nervous system disorders) | 0 | 1 | 1 | 1
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Acute febrile illness (General disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zinc and Probiotic (N=154) | Zinc Alone (N=155) | Probiotic Alone (N=154) | Placebo (N=155)
Diarrhea (Gastrointestinal disorders) | 38 | 47 | 44 | 31
Vomiting (Gastrointestinal disorders) | 29 | 29 | 32 | 33
Fever (General disorders) | 112 | 117 | 108 | 100
Cough (Respiratory, thoracic and mediastinal disorders) | 130 | 134 | 128 | 130
Cold/runny nose (Respiratory, thoracic and mediastinal disorders) | 143 | 148 | 140 | 144
Any other illness (General disorders) | 31 | 34 | 37 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No